CLINICAL TRIAL: NCT02491593
Title: Quantitative Immunochemical Fecal Occult Blood Test in Symptomatic Patients
Acronym: FIKA
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: QFecalBlood 2013/2:7
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Neoplasms
Keywords: fecal occult blood
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: fecal occult blood test

SUMMARY:
The aim of this study is to compare the outcome of three (3) quantitative immunochemical faecal occult blood test in symptomatic patients.

DETAILED DESCRIPTION:
Consecutive patients referred from primary care for colonoscopy due to symptoms are eligible. Patients will receive written information of the study together with the time for colonoscopy. A specific research nurse will call them and for those accepting participation, history and current medication will be collected. Kits will be sent to patients and they will provide three faecal samples before examination. These will be analysed at one certified laboratory.

Hemoglobin concentration will be notified in the range of 50 - < 1000 ng/mL, or as a negative outcome.

Macroscopic findings at the colonoscopy will be collected, as well as the outcome of the pathological report.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms associated with colorectal cancer (anemia, change of bowel habits, diarrhoea, constipation, haematochezia, weight loss, anorexia)

Exclusion Criteria:

* Screening investigations
* High-risk patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred from primary care for investigation of symptoms potentially caused by colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with high fecal blood output in relation to colorectal cancer | Up to 36 months
  Accuracy of diagnosis in colorectal cancer

SECONDARY OUTCOMES:
Number of patients with low fecal blood output in relation to colorectal polyps | Up to 36 months
  Accuracy of diagnosis of colorectal polyps

CONTACTS AND LOCATIONS:
Overall Officials: Louise Olsson, MD, PhD, Principal Investigator — Centre for Clinical research, Eskilstuna, Uppsala universitet
Locations (1):
- Unit of Endoscopy, Eskilstuna, Sweden

REFERENCES:
- [Derived] Tsapournas G, Hellstrom PM, Cao Y, Olsson LI. Diagnostic accuracy of a quantitative faecal immunochemical test vs. symptoms suspected for colorectal cancer in patients referred for colonoscopy. Scand J Gastroenterol. 2020 Feb;55(2):184-192. doi: 10.1080/00365521.2019.1708965. Epub 2020 Jan 6. PMID 31906738